CLINICAL TRIAL: NCT00027053
Title: Trazodone for Sleep Disturbance - Early Alcohol Recovery
Brief Title: Trazodone for Sleep Disturbance in Early Alcohol Recovery
Acronym: SIESTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Peter Friedmann, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAAFRI13243; R01AA013243 (NIH); NIH grant R01 AA013243
Record Dates: First submitted 2001-11-19; First posted 2001-11-20 (Estimated); Last update posted 2010-05-13 (Estimated); Status verified 2006-03

CONDITIONS: Alcoholism
Keywords: alcoholism; alcohol dependence; trazadone; sleep
MeSH Terms: conditions — Alcoholism | interventions — Trazodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trazodone (Experimental)
  Interventions: Drug: Trazodone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trazodone — 50 to 150 mg qhs
  Arms: Trazodone
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind clinical trial comparing trazodone (Desyrel) and placebo among sleep-disturbed, alcohol-dependent individuals shortly after discharge from an inpatient detoxification program. Subjects will undergo a baseline assessment and random assignment to trazodone or identical placebo for 12 weeks. All persons completing the alcohol detoxification at Stanley Street Treatment and Resources (SSTAR) will be screened. (SSTAR of Rhode Island provides detoxification services to non/underinsured persons of Rhode Island.)

ELIGIBILITY:
Inclusion Criteria:

* Completed an alcohol detoxification program.
* Meets criteria for alcohol dependence.
* Meets criteria for sleep disturbance.
* If female of childbearing potential must be using adequate contraception.
* Has a location to which they will return after the initial research interview and a person they regularly contact.
* Speaks English sufficiently to understand instructions and assessment.

Exclusion Criteria:

* Meets criteria for substance dependence for sedative/hypnotic drugs, stimulants, cocaine or opiates, or of organic brain disorder, bipolar disorder, schizophrenia, schizoaffective, schizophreniform, or paranoid disorder, or major depression.
* Current suicidality.
* Use of psychotropic, antidepressant, anxiolytic or antidipsogenic medication.
* Inability or refusal to terminate the use of proerectile agents, herbal medications or sleep medication for the study period.
* The presence of contraindications to the study medications, including pregnancy/lactation, ischemic heart disease, cardiac arrhythmias, priapism or hypotension.
* Presence of comorbid medical conditions associated with sleep disturbance including obstructive sleep apnea, poorly controlled diabetes mellitus or emphysema.
* Evidence of neuropsychological dysfunction.
* Probation/parole requirements that might interfere with participation in study.
* Inability to identify at least one contact person.
* Living on the street after detoxification (homeless persons living in a shelter, halfway house or other residence will not be excluded).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2002-06; Primary Completion 2006-01 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Percent days abstinent from alcohol (PDA) | 12 and 24 weeks

SECONDARY OUTCOMES:
sleep quality | 12 and 24 weeks
Drinks per drinking day | 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter D. Friedmann, MD, MPH, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Result] Friedmann PD, Rose JS, Swift R, Stout RL, Millman RP, Stein MD. Trazodone for sleep disturbance after alcohol detoxification: a double-blind, placebo-controlled trial. Alcohol Clin Exp Res. 2008 Sep;32(9):1652-60. doi: 10.1111/j.1530-0277.2008.00742.x. Epub 2008 Jul 8. PMID 18616688